CLINICAL TRIAL: NCT07160348
Title: Translation and Validation of the Hypoparathyroidism Patient Experience Scales (HPES) Questionnaire in Patients With Hypoparathyroidism for Use in the Greek Population
Brief Title: Translation and Validation of the Hypoparathyroidism Patient Experience Scales (HPES) Questionnaire in Greek
Acronym: HPES
Status: Not yet recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: National and Kapodistrian University of Athens (Other); 424 General Military Hospital (Other); General Hospital Of Thessaloniki Ippokratio (Other); Laikο General Hospital, Athens (Other); 251 Hellenic Air Force & VA General Hospital (Other); Hellenic Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Panagiotis Anagnostis, Assistant Professor, Aristotle University Of Thessaloniki
Other Study IDs: 8802
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hypoparathyroidism
Keywords: hypoparathyroidism; parathyroid hormone; palopegteriparatide; calcium metabolism disorders
MeSH Terms: conditions — Hypoparathyroidism; Calcium Metabolism Disorders | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with chronic hypoparathyroidism: Patients ≥18 years of age, fluent in Greek language, diagnosed with chronic hypoparathyroidism (HP), on optimal treatment with calcium and active vitamin D metabolites. Chronic HP is defined when continuous therapy with calcium and vitamin D is required for >12 months.
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Translation and validation of the existing HPES-Symptom and HPES-Impact Questionnaires in the Greek population

SUMMARY:
This is a crossectional study that will be conducted at several tertiary centers in Greece.

To participate in the study, patients should be ≥18 years of age, fluent in Greek language, diagnosed with chronic HP, on optimal treatment with calcium and active vitamin D metabolites. Chronic HP is defined when continuous therapy with calcium and vitamin D is required for >12 months.

Exclusion criteria will include:

1. Patients inadequately controlled with conventional therapy:

   1. corrected serum Ca (cCa) ≤8 mg/dl or cCa ≤8.2 mg/dl with symptoms of hypocalcemia
   2. serum P >5.5 mg/dl
2. Age >80 years
3. Presence of neoplastic disease
4. Pregnancy
5. Diagnosis of psychiatric disease or cognitive impairment
6. Participants experiencing other comorbidities that may affect QoL
7. Lack of informed consent The study will seek approval from the Ethics in Research Committee of its participating center. All participants will be informed about the objectives of the study and will sign an informed consent.

The HPES-Symptom was developed in accordance with the Food and Drug Administration guidance and best research practices for PRO measure development. The methodology used has been previously described.

The first step of the translation process requires two forward translations of the English version of the questionnaire. The translations will be done by two translators who are native speakers of the target (Greek) language and can understand the English version. Then a reconciled translation is made based on the two translations - that is, the chief investigator will review the two translations to achieve the best possible version by choosing one of the two translations or by combining them on the basis of their correctness, wording etc.

The next step requires translating the reconciled version back into English, again done by two translators who will be native speakers of English or at least will have a very good command of English.

DETAILED DESCRIPTION:
1. Background Hypoparathyroidism (HP) is a chronic disease, characterized by hypocalcemia and hyperphosphatemia, due to low, or inappropriately normal, concentrations of parathyroid hormone (PTH). It is usually the result of remnant parathyroid tissue dysfunction, after thyroidectomy or parathyroidectomy. It is rarely due to autoimmune or genetic disorders. In contrast to other endocrine diseases, patients with HP are typically managed with conventional therapy, which includes oral calcium and active vitamin D. In patients with chronic HP who are refractory or experience intolerance to conventional therapy, replacement therapy with PTH should be considered. Despite the achievement of normal serum calcium and phosphate levels, HP may be associated with increased risk of chronic complications, such as basal ganglia calcification, cataract, nephrolithiasis, chronic kidney disease (CKD), neuropsychiatric disorders and increased mortality.

   Another underestimated issue in patients with HP is impairment of quality of life (QoL) in comparison with healthy controls, as well as with patients with a history of thyroidectomy. So far, several scales to assess clinical symptoms and QoL in HP have been used, such as the Short Form-36 (SF-36, although non-specific), as well the disease-specific Hypoparathyroid Patient Questionnaire (HPQ 40/28) and the Hypoparathyroidism Patient Experience Scales (HPES), including the 17-item HPES-Symptom and the 26-item HPES-Impact tools. However, these disease-specific QoL questionnaires have not yet been translated and validated into the Greek language for patients with HP, which is essential for culturally relevant data collection and improved clinical care in this population.

   The aim of the present study is to translate and validate the HPES-Symptom and the HPES-Impact questionnaires for patients with HP for use in the Greek population.
2. Study methodology

2.1 Subjects and Settings This is a cross-sectional study that will be conducted at several tertiary centers in Greece.

To participate in the study, patients should be ≥18 years of age, fluent in Greek language, diagnosed with chronic HP, on optimal treatment with calcium and active vitamin D metabolites. Chronic HP is defined when continuous therapy with calcium and vitamin D is required for >12 months.

Exclusion criteria will include:

1. Patients inadequately controlled with conventional therapy:

   1. corrected serum Ca (cCa) ≤8 mg/dl or cCa ≤8.2 mg/dl with symptoms of hypocalcemia
   2. serum P >5.5 mg/dl
2. Age >80 years
3. Presence of neoplastic disease
4. Pregnancy
5. Diagnosis of psychiatric disease or cognitive impairment
6. Participants experiencing other comorbidities that may affect QoL
7. Lack of informed consent The study will seek approval from the Ethics in Research Committee of its participating center. All participants will be informed about the objectives of the study and will sign an informed consent.

2.2 Design and Instruments 2.2.1 HPES - Symptom and HPES - Impact Questionnaires HPES - Symptom The HPES-Symptom was developed in accordance with the Food and Drug Administration guidance and best research practices for PRO measure development. The methodology used has been previously described. HPES-Symptom measure includes 17 items across two domains of signs and symptoms: Physical and Cognitive. Response options are based on a five-point Likert-type scale, chosen to ensure that meaningful distinctions could be made among responses for analysis while minimizing the cognitive burden for respondents completing the instrument. Response options included "Never", "Occasionally (1-25% of the time)", "Sometimes (26-50% of the time)", "Often (51-75% of the time)", and "Very Often/Always (76-100% of the time)".

HPES - Impact The HPES-Impact was developed in accordance with the FDA guidance on best research practices for PRO measure development. The methods used to carry out this research, including eligibility criteria, have been described in detail in the HPES-Symptom article. HPES-Impact measure includes 26 items across four domains of QOL: Physical Functioning, Daily Life, Psychological Well-Being, and Social Life and Relationships. Response options are based on a 5-point Likert-type scale (response options: "Not at all," "A little," "Moderately," "A lot," and "Extremely").

2.2.2 Translation Process The first step of the translation process requires two forward translations of the English version of the questionnaire. The translations will be done by two translators who are native speakers of the target (Greek) language and can understand the English version. Then a reconciled translation is made based on the two translations - that is, the chief investigator will review the two translations to achieve the best possible version by choosing one of the two translations or by combining them on the basis of their correctness, wording etc.

The next step requires translating the reconciled version back into English, again done by two translators who will be native speakers of English or at least will have a very good command of English.

2.2.3 Pilot Testing Once the translation process is completed, the final document can undergo linguistic validation, the so-called pilot-testing. It includes a group of 30-40 patients, who comment on the comprehensibility of the translation. All the comments obtained by the pilot testing phase will be reviewed and if relevant will be incorporated in the final version of the translation.

All patients should be native speakers of the target language and constitute a representative group in terms of socio-demographic characteristics (gender, age and education).

The pilot testing step consists of two parts:

1. Patients receive the translated questionnaire and fill it in.
2. A researcher discusses the translation with the patients individually or in a focus group setting.

If any items elicited comments because of problems with comprehensibility and the chief investigator suggests a change in the wording, the item has to be re-tested on a few patients, including the patients that reported the comprehension problems and some that did not report any problems. The re-test serves to ensure that the problem has been solved and that the new version is understandable for everybody. In the re-test the interviewer will only check the problematic items with the patients and not the whole questionnaire.

2.3 Sociodemographic Data

The sociodemographic characteristics of each patient will be captured. More specifically these will include:

1. Name, age, gender
2. Marital status
3. Occupations
4. Education
5. Height, weight, body mass index, blood pressure, heart rate
6. Etiology of HP (Post Surgical vs. Non-surgical)
7. Type of surgery (thyroidectomy, parathyroidectomy)
8. Duration of HP
9. Reason for operation (thyroid Cancer, Graves' disease, multinodular goiter, primary hyperparathyroidism (adenoma vs. parathyroid gland hyperplasia)
10. Co-morbidities
11. History of fractures and falls
12. Total daily dose of calcium, active vitamin D and cholecalciferol
13. Thiazide diuretic use
14. Other concomitant medications
15. Calcium metabolism [serum total calcium (Ca), albumin, phosphate (P), magnesium, creatinine, as well as 24h-urinary calcium, creatinine and sodium]
16. Hormonal profile, including thyroid stimulating hormone, PTH, 25-hydroxy-vitamin D
17. Fasting blood glucose, aspartate transaminase, alanine transaminase, alkaline phosphatase, lipid profile
18. Kidney ultrasound
19. Bone mineral density in lumbar spine, femoral neck and total hip

2.4 Statistical Analysis Statistical analyses will be performed to establish the reliability and the validity of the Greek questionnaire. Evaluation of reliability will be based on the internal consistency analysis through Cronbach's alpha coefficient.

A construct and convergent validity will be performed via comparing the HPES questionnaires with a generic QoL instrument, the SF-36. The level of significance is set at p≤0.05.

To reduce responses bias, subjects will also be asked to rate their overall health and overall QOL on 100-point scales (higher scores indicating greater satisfaction).

3. Timeline

* Months 0-2: translation process
* Months 3-6: recruitment and data collection
* Months 7-8: data analysis
* Months 8-12: final report writing and dissemination of results

ELIGIBILITY:
Inclusion Criteria:

Patients should be ≥18 years of age, fluent in Greek language, diagnosed with chronic HP, on optimal treatment with calcium and active vitamin D metabolites. Chronic HP is defined when continuous therapy with calcium and vitamin D is required for >12 months.

Exclusion Criteria:

1. Patients inadequately controlled with conventional therapy:

   1. corrected serum Ca (cCa) ≤8 mg/dl or cCa ≤8.2 mg/dl with symptoms of hypocalcemia
   2. serum P >5.5 mg/dl
2. Age >80 years
3. Presence of neoplastic disease
4. Pregnancy
5. Diagnosis of psychiatric disease or cognitive impairment
6. Participants experiencing other comorbidities that may affect QoL
7. Lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hypoparathyroidism ≥18 years of age
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Translation and validation the HPES-Symptom and the HPES-Impact questionnaires in Greek | 6 months
  To translate and validate the HPES-Symptom and the HPES-Impact questionnaires for patients with chronic hypoparathyroidism for use in the Greek population
Translation and validation the HPES-Symptom and the HPES-Impact questionnaires in Greek | 12 months
  To translate and validate the HPES-Symptom and the HPES-Impact questionnaires for patients with chronic hypoparathyroidism for use in the Greek population

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khan AA, Rejnmark L, Rubin M, Schwarz P, Vokes T, Clarke B, Ahmed I, Hofbauer L, Marcocci C, Pagotto U, Palermo A, Eriksen E, Brod M, Markova D, Smith A, Pihl S, Mourya S, Karpf DB, Shu AD. PaTH Forward: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial of TransCon PTH in Adult Hypoparathyroidism. J Clin Endocrinol Metab. 2022 Jan 1;107(1):e372-e385. doi: 10.1210/clinem/dgab577. PMID 34347093
- [Background] Khan AA, Bilezikian JP, Brandi ML, Clarke BL, Gittoes NJ, Pasieka JL, Rejnmark L, Shoback DM, Potts JT, Guyatt GH, Mannstadt M. Evaluation and Management of Hypoparathyroidism Summary Statement and Guidelines from the Second International Workshop. J Bone Miner Res. 2022 Dec;37(12):2568-2585. doi: 10.1002/jbmr.4691. Epub 2022 Nov 14. PMID 36054621